CLINICAL TRIAL: NCT00000888
Title: A Phase I Trial of the Safety, Tolerance, and Pharmacokinetics of Oral Ritonavir Co-Administered With Lamivudine (3TC) and Zidovudine (ZDV) in HIV-1-Infected Pregnant Women and Their Infants
Brief Title: Safety and Effectiveness of Ritonavir Plus Lamivudine Plus Zidovudine in HIV-Infected Pregnant Women and Their Babies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 354; 10604 (Registry Identifier: DAIDS ES); PACTG 354
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Drug Therapy, Combination; Administration, Oral; Zidovudine; HIV Protease Inhibitors; Ritonavir; Disease Transmission, Vertical; Anti-HIV Agents; Fetal Blood
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — Ritonavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give ritonavir (RTV) plus lamivudine (3TC) plus zidovudine (ZDV) to HIV-infected pregnant women during pregnancy and to their babies after birth.

Pregnant women who are HIV-positive are at risk of giving HIV to their babies during pregnancy or delivery. It is important to learn how to prevent HIV-positive pregnant women from giving HIV to their babies. RTV and ZDV have been shown to be safe and effective against HIV in adults. The combination of 3 anti-HIV drugs (RTV, 3TC, and ZDV) may help prevent HIV infection from mother to infant but studies are needed to determine whether they are safe and effective during pregnancy.

DETAILED DESCRIPTION:
Controlled studies of the pharmacokinetics and safety of new drugs are critical to the development of alternative therapies for the prevention of perinatal transmission of HIV-1. The dosing regimen of RTV and ZDV used to treat pregnant women in this study has been shown to be safe and effective against HIV in adults. Little is known about the metabolism and tolerance of these drugs during pregnancy, and Phase I studies are needed to determine dosage, safety, and tolerance. Protease inhibitors in combination with other antiretroviral drugs may help reduce the rate of perinatal transmission of HIV-1.

Pregnant women start with RTV (increasing gradually over a few days) plus 3TC plus ZDV until active labor. Intrapartum, women receive RTV plus 3TC plus ZDV, then postpartum (after cord clamped until 12 weeks postpartum), RTV plus 3TC plus ZDV. [AS PER AMENDMENT 2/9/99: For maternal dosing, one Combivir tablet (containing 3TC and ZDV) may be administered in place of the individual agents 3TC and ZDV. During the intrapartum period, Combivir is held and the patient follows intrapartum 3TC/ZDV dosing. During the intrapartum period, no RTV is given after the onset of active labor. During the postpartum period, RTV is begun as soon as oral intake is allowable following delivery. During the postpartum period, Combivir may be resumed. All subjects who prematurely discontinue study treatment should continue to be followed for the duration of the study.] [AS PER AMENDMENT 9/28/99: During the intrapartum period, RTV is given at the start of active labor.] Infants begin 3TC and ZDV as soon as oral intake is tolerated. Infants participate in one of two cohorts. The first four infants delivered (Cohort 1) receive RTV as a single dose between Days 8 and 12. The next six infants delivered (Cohort 2) start RTV at 2-3 days of life. The dosing schedule is based on Cohort 1 drug pharmacokinetics data. [AS PER AMENDMENT 2/9/99: Cohort 1 is expanded to seven mother/infant pairs.] [AS PER AMENDMENT 9/28/99: Cohort 1 is expanded to eight mother/infant pairs.] Both maternal and infant blood is drawn to assess drug pharmacokinetics. Cervical secretions are collected to assess presence of virus. In addition, all placentas are examined by histopathology to determine the role of placenta on preterm delivery in women receiving combination antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria

Women may be eligible for this study if they:

* Are HIV-positive.
* Are between 14 and 32 weeks pregnant.
* Are at least 13 years old (consent of parent or guardian required if under 18).
* Have the consent of the baby's father (if he can be reached).

Exclusion Criteria

Women will not be eligible for this study if they:

* Are having problems with their pregnancy.
* Have a history of problem pregnancies including miscarriages, birth defects, stillbirths, or giving birth to premature or low-birth-weight babies.
* Have had side effects to ZDV, 3TC, or RTV.
* Have an active opportunistic (AIDS-related) or other serious infection.
* Have other serious conditions such as heart or lung problems, blood disorders, diabetes, or seizures.
* Are pregnant with more than one baby (such as twins or triplets).
* Are taking other experimental medications.
* Are taking other anti-HIV medications.
* Are taking certain other medications including those for cancer, blood pressure, or seizures.
* Are abusing drugs or alcohol.
* Are breast-feeding.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14
Dates: Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Scott, Study Chair — Univ of Miami (Pediatric); Mary Jo O'Sullivan, Study Chair — Univ of Miami (Pediatric)
Locations (5):
- United States (5):
  - Univ. of Miami Miller School of Medicine - Jackson Memorial Hosp., Miami, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - St. Jude/UTHSC CRS, Memphis, Tennessee

REFERENCES:
- [Result] Chadwick EG, Rodman JH, Britto P, Powell C, Palumbo P, Luzuriaga K, Hughes M, Abrams EJ, Flynn PM, Borkowsky W, Yogev R; PACTG Protocol 345 Team. Ritonavir-based highly active antiretroviral therapy in human immunodeficiency virus type 1-infected infants younger than 24 months of age. Pediatr Infect Dis J. 2005 Sep;24(9):793-800. doi: 10.1097/01.inf.0000177281.93658.df. PMID 16148846